CLINICAL TRIAL: NCT06323733
Title: Exercise Intervention for Patients With Cancer Cachexia: Effects of a 12-week Supervised Program and One-year Follow-up of Patients and Cachexia-related Symptoms
Brief Title: Exercise Intervention for Patients With Cancer Cachexia: Effects of a 12-week Program and One-year Follow-up.
Acronym: 2CAPA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Peyrachon Romane (Other)
Responsible Party: Sponsor-Investigator, Peyrachon Romane, Investigator, PhD, University of Rennes 2
Organization: University of Rennes 2 (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2CAPA
Record Dates: First submitted 2024-03-08; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Cachexia-Anorexia Syndrome
Keywords: Cachexia; Cancer; Exercise; Body composition; Quality of life
MeSH Terms: conditions — Cachexia; Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise intervention (Experimental): The exercise intervention will consist of a personalized and supervised program lasting 12 weeks with two sessions per week, held on Tuesdays and Thursdays at the Sports and Medicine Center SPORMED in Rennes, France.
  Each session will combine endurance and resistance training, commencing with a 6-minute cardiovascular warm-up on ergometers (cycling ergometer or treadmill). This will be followed by 20 minutes at moderate intensity (60-70% of Heart Rate Reserve (HRR)), concluding with a 2-minute recovery period at light intensity. Heart rate will be monitored using a pulse oximeter. Participants will report their rate of perceived exertion during endurance training using a 5-point scale ("very easy," "easy," "moderate," "difficult," "very difficult").
  Interventions: Other: Exercise Intervention

INTERVENTIONS:
Other: Exercise Intervention — The exercise intervention will consist of a personalized and supervised program lasting 12 weeks with two sessions per week, held on Tuesdays and Thursdays at the Sports and Medicine Center SPORMED in Rennes, France. Each session will last 1 hour under the supervision of physiotherapists. Each session will combine endurance and resistance training, commencing with a 6-minute cardiovascular warm-up on ergometers (cycling ergometer or treadmill). This will be followed by 20 minutes at moderate intensity (60-70% of

SUMMARY:
The prevalence of cancer with cachexia is rising sharply. More than 80% of digestive cancer patients are affected by cancer cachexia. Cachexia leads to weight loss, and reduces quality of life (QoL), cancer treatment response and survival. Exercise could counteract the deleterious effects of cachexia. The 2CAPA study aims to assess the effectiveness of a 12-week exercise program on various symptoms associated with cancer cachexia, including Health-Related QoL (HRQoL), fatigue, appetite, body composition, physical fitness, and physical activity levels. Additionally, it seeks to examine compliance with the exercise program, identify barriers to regular exercise and determine how compliance influences physical and psychological effects. Furthermore, this study aims to determine the maintenance of physical activity levels and the effects post-program for one year follow-up on cachexia-related symptoms.

Methods: This study will include 31 cancer patients with cachexia. Participants will receive a supervised exercise program lasting 12-weeks with two sessions per week combining endurance and resistance training. Outcomes include HRQoL, fatigue, appetite, anthropometric parameters, physical performances, and physical activity levels at baseline, at the end of the 12-week exercise program, and at 3-, 6- and 12- months post-intervention.

DETAILED DESCRIPTION:
Study objectives and design:

The 2CAPA study will aim to assess the efficacy of a supervised 12-week APA program on cachexia symptoms; HRQoL (global QoL, fatigue, physical functioning, appetite, and pain), cancer-related fatigue, appetite, body composition (weight, lean mass, fat mass), appetite, physical condition (endurance, strength, balance), and physical activity and sedentary levels. The secondary aim will be to assess the compliance to exercise program and barriers that could affect compliance, and to explore how compliance may impact the magnitude of the observed effects. The third objective will be to determine the maintenance of physical activity levels and the effects of exercise for 1 year follow-up (at the 3-months, 6-months and 12-mon

ths follow-ups assessments) on cachexia symptoms. In summary, this study aims to assess the effectiveness of a 12-week exercise program on various parameters affected by cancer-related cachexia and identify barriers to regular participation to exercise program. Patient behavior and outcomes will then be assessed during a one-year post-program follow-up.

The 2CAPA study is a prospective, single-arm study conducted in a sport and medicine center. The study is promoted by the University of Rennes 2 (Rennes, France).

Recruitment:

Patients can join the program spontaneously or after receiving information at the hospital. At the hospital, patients diagnosed with cancer cachexia will undergo eligibility screening by clinicians within the Digestive Tract Diseases department of Rennes University Hospital (CHU Rennes, France). Clinicians will identify suitable participants and refer them to the sports-medical center SPORMED (Rennes, France), located outside the hospital, where the sessions will take place. A practice setting outside the hospital can encourage engagement and enable the study of the effects of exercise by being as close as possible to people's real-life conditions. The physiotherapist at the sports-medical center will provide participants with information about the possibility and benefits of exercise. Additionally, the physiotherapist will guide patients to the sports-medical center SPORMED (Rennes, France), where the sessions will take place. Patients enrolled in the exercise program will then receive both oral and written information about the trial. All participants will be required to sign and provide an informed consent form.

Intervention :

Exercise intervention:

The exercise intervention will consist of a personalized and supervised program lasting 12 weeks with two sessions per week, held on Tuesdays and Thursdays at the Sports and Medicine Center SPORMED in Rennes, France. Patients will have the flexibility to choose their session time between 11:30 a.m. and 4 p.m and each session will last 1 hour under the supervision of physiotherapists. The program will include both aerobic and resistance exercises. The program will adhere to the principle of "autoregulation," allowing for a reduction in exercise intensity and/or duration when treatment-related side effects will be heightened. Patients will be encouraged to maintain the prescribed exercise intensity and duration if treatment-related side effects will be manageable.

Each session will combine endurance and resistance training, commencing with a 6-minute cardiovascular warm-up on ergometers (cycling ergometer or treadmill). This will be followed by 20 minutes at moderate intensity (60-70% of Heart Rate Reserve (HRR)), concluding with a 2-minute recovery period at light intensity. Heart rate will be monitored using a pulse oximeter. Participants will report their rate of perceived exertion during endurance training using a 5-point scale ("very easy," "easy," "moderate," "difficult," "very difficult"). Session intensity will be determined based on the HRR, which will be calculated with the theoretical maximal heart rate (HR maximal) and resting heart rate (HR rest) of the patient, with adjustments made according to the patient's feedback and treatment-related side effects.

Subsequently, resistance training will begin with a mobility warm-up, followed by exercises involving body weight, free weight, elastics, swissball, etc. The protocol for resistance training is described in the Supplemental Material. Patients will perform 2 to 4 sets per exercise and 8 to 14 repetitions.

Outcomes will be assessed at baseline (at the initiation of the program), post-intervention (at the end of the program), and at 3, 6, and 12 months of follow-up. All assessments will be conducted by an exercise physiologist. Demographics and treatment and diagnosis characteristics were collected at baseline during a short interview.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of cancer cachexia according to Martin's classification
* Undergoing treatment or within 1 year post-treatment (of any type), with or without metastasis
* Eastern Cooperative Oncology Group Performance status ≤ 2, 5) life expectancy ≥ 3 months
* Willingness to actively participate throughout the study
* Ability to engage in supervised exercise program as certified by their oncologist
* Valid health insurance affiliation,
* Proficiency in reading, writing, and understanding French.

Exclusion Criteria:

* Exhibit central nervous system involvement with neurological deficits restricting walking
* Are concurrently participating in another exercise intervention study,
* Are pregnant
* Are under legal or administrative detention/ deprived of liberty by judicial or administrative decision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Health-Related Quality of Life | Through study completion : Baseline, 12 weeks, 24 weeks, 36 weeks, 60 weeks
  Health-Related Quality of Life: The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) version 3.0 will be used to assess changes in levels of health-related Quality of Life (QOL). The EORTC QLQ-C30 is an internationally validated, concise, self-reporting cancer-specific measure of health-related QOL (25). This scale comprises 30 items, including one global health status/QOL scale and five multi-item functional scales evaluating physical, role, emotional, cognitive, and social function. Additionally, three multi-item symptom scales assess fatigue, pain, and nausea/vomiting, and six single items assess symptoms such as dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties. A high score for the global health status and QoL and for the functional scales represents a high level of QoL and functioning. Nevertheless, a high score for a symptom scale / item represents a high level of symptomatology.

SECONDARY OUTCOMES:
Body weight | Through study completion : Baseline, 12 weeks, 24 weeks, 36 weeks, 60 weeks
  Body weight (in kilograms) will be measured by bioelectrical impedance analysis (Tanita, DC-360).
Body mass index | Through study completion : Baseline, 12 weeks, 24 weeks, 36 weeks, 60 weeks
  Weight (in kilograms) and height (in meters) will be combined to report BMI in kg/m^2
Lean mass | Through study completion : Baseline, 12 weeks, 24 weeks, 36 weeks, 60 weeks
  Lean mass (in kilograms and expressed as a percentage of total body weight will be determined by bioelectrical impedance analysis (Tanita, DC-360).
Fat mass | Through study completion : Baseline, 12 weeks, 24 weeks, 36 weeks, 60 weeks
  Fat mass (in kilograms and expressed as a percentage of total body weight) will be determined by bioelectrical impedance analysis (Tanita, DC-360).
Aerobic fitness | Through study completion : Baseline, 12 weeks, 24 weeks, 36 weeks, 60 weeks
  Aerobic fitness: Participants will undergo a 6-minute walk test on a flat, indoor, 20-meter walkway.
Muscular strength of the lower limbs | Through study completion : Baseline, 12 weeks, 24 weeks, 36 weeks, 60 weeks
  Muscular strength of the lower limbs will be assessed using the sit-to-stand (30 seconds) test.
Handgrip strength | Through study completion : Baseline, 12 weeks, 24 weeks, 36 weeks, 60 weeks
  The muscular strength of the upper limbs will be assessed through a handgrip test using a hand dynamometer (Takei 5401 Hand Grip Dynamometer (digital)) and expressed in kilograms.
Static balance ability | Through study completion : Baseline, 12 weeks, 24 weeks, 36 weeks, 60 weeks
  Static balance ability will be assessed using a one-leg stand test, performances will be expressed in seconds.
Appetite | Through study completion : Baseline, 12 weeks, 24 weeks, 36 weeks, 60 weeks
  Appetite will be assessed using the SEFI (Simple Evaluation of Food Intake). SEFI is a scale that evaluates the quantity of ingesta from 1 to 10. A score of 7 or less indicates anorexia
Cancer-related Fatigue | At baseline and at 12 weeks
  Fatigue will be measured using the Multidimensional Fatigue Inventory (MFI-20). The questionnaire consists of 20 statements in which the patient rate themselves on a Likert scale ranging from 1 ("strongly disagree") to 5 ("strongly agree")
Physical Activity and Sedentary Levels | Through study completion : Baseline, 12 weeks, 24 weeks, 36 weeks, 60 weeks
  Participants will recall and self-report their physical activity levels (frequency and duration of vigorous intensity, moderate intensity, walking, and sitting) during the previous 7 days, using the International Physical Activity Questionnaire Short Form (IPAQ-SF). Depending on their results, patients may be considered sedentary, inactive, moderately active or very active.
Stages of change for exercise | Through study completion : Baseline, 12 weeks, 24 weeks, 36 weeks, 60 weeks
  The stages of change for exercise will be evaluated by a scale derived from the transtheoretical model of behavior change.
Exercise beliefs | At baseline and at 12 weeks
  Exercise beliefs will be assessed through the Cancer Exercise Stereotypes Scale (CESS). The questionnaire consists of 19 statements in which the patients rate themselves on a Likert scale ranging from 1 ("strongly disagree") to 6 ("strongly agree").

OTHER OUTCOMES:
Compliance to exercise intervention | During the 12-week program
  The overall compliance rate will be calculated as the number of completed exercise sessions/total prescribed sessions.
Reasons for absence | During the 12-week program
  Reasons for missed sessions will be collected from the participant by phone or at their next session. Reasons will be categorized into medical reasons, personal reasons, environmental reasons, and professional reasons.
Timing of absences | During the 12-week program
  The timing of absences will also be recorded and studied. The timing of absences will be expressed in the form start of program, middle of program, end of program
Fidelity to session duration | During the 12-week program
  Fidelity rates will be determined by comparing the prescribed duration of session versus actual exercise duration (in minutes)
Fidelity to session intensity | During the 12-week program
  Intensity fidelity rates will be determined by comparing the prescribed intensity versus actual exercise intensity (expressed in percentage of Heart-Rate Reserve and self-perception of effort).
Reasons to modify exercise sessions | During the 12-week program
  The occurrence and reasons for adjustments in aerobic exercise intensity will be recorded by a physiotherapist.
Incidence of Adverse Events | During the 12-week program
  Physiotherapists will monitor and record serious adverse events and program interruptions due to exercise complications.

CONTACTS AND LOCATIONS:
Overall Officials: Romane Peyrachon, MhD, Principal Investigator — Rennes 2 University, M2S lab EA7470; Amélie Rébillard, PhD, Study Director — Rennes 2 University, M2S lab EA7470
Locations (1):
- SPORMED, Rennes, Brittany Region, France

IPD SHARING:
Plan to Share IPD: Yes
The study protocol will be published. Anonymized patient data and statistical analyses will be available.
Supporting Information: Study Protocol, ICF
Time Frame: Information will be available in 2024 for an infinite duration.
Access Criteria: Open access

REFERENCES:
- [Derived] Peyrachon R, Richard C, Gelein B, Lievre A, Andre N, Chaory K, Rebillard A. Rationale and design of an exercise intervention for patients with cancer cachexia: protocol for a one-year follow-up prospective study (2CAPA). BMC Sports Sci Med Rehabil. 2025 May 24;17(1):129. doi: 10.1186/s13102-025-01173-8. PMID 40413464